CLINICAL TRIAL: NCT04044209
Title: A Phase II of the IDH1 Inhibitor AG-120 in Combination With the Checkpoint Blockade Inhibitor, Nivolumab, for Patients With IDH1 Mutated Relapsed/Refractory AML and High Risk MDS
Brief Title: A Study of the IDH1 Inhibitor AG-120 in Combination With the Checkpoint Blockade Inhibitor, Nivolumab, for Patients With IDH1 Mutated Relapsed/Refractory AML and High Risk MDS
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients were able to be screened nor enrolled.
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000024263
Record Dates: First submitted 2019-07-25; First posted 2019-08-05 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Myelodysplastic Syndromes; Acute Myeloid Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myeloid, Acute | interventions — ivosidenib; Nivolumab

STUDY DESIGN:
Intervention Model Description: The study is a single arm phase II trial with a safety cohort
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Patients receiving nivolumab and ivosidenib (Experimental): Patients who meet eligibility criteria will initiate therapy with the IDH1 inhibitor ivosidenib (AG-120) that will be administered orally on a continuous basis at the dose of 500 mg/day starting at day 1 of each cycle. A cycle will be defined as a 28-day period.
  On Cycle 2 day 1 the patient will receive nivolumab 480mg once. This will be repeated on Day 1 of every subsequent cycle. Patient will be treated until progression, transplant or unacceptable toxicity. The patient will be continually monitored on therapy and will undergo scheduled response assessments to evaluate response.
  Interventions: Drug: AG-120; Drug: Nivolumab

INTERVENTIONS:
Drug: AG-120 — The IDH1 inhibitor ivosidenib (AG-120) that will be administered orally on a continuous basis at the dose of 500 mg/day starting at day 1 of each cycle. A cycle will be defined as a 28-day period.
Drug: Nivolumab — On Cycle 2 day 1 the patient will receive nivolumab 480mg once. This will be repeated on Day 1 of every subsequent cycle.

SUMMARY:
In this trial the investigators aim to evaluate safety and efficacy of combination Ivosidenib (AG-120) and nivolumab in the context of adult patients with Isocitrate dehydrogenase-1 (IDH1) mutated acute myeloid leukemias (AML) or Myelodysplastic syndromes (MDS).

DETAILED DESCRIPTION:
Primary objectives:

1. To determine the overall response rate of (CR/CRi) of combination ivosidenib (AG-120) and nivolumab in patients with high risk MDS and relapsed/ refractory AML
2. To determine the duration of response of combination ivosidenib (AG-120) and nivolumab in patients with high risk MDS and relapsed/ refractory AML 2.2 Secondary Objectives

1) To determine the progression free survival of patients treated with combination ivosidenib (AG- 120) and nivolumab. 2) To determine the overall survival of patients treated with combination ivosidenib (AG-120) and nivolumab. 3) To determine hematological response rate of patients treated with combination ivosidenib (AG- 120) and nivolumab. 4) To establish the duration of response to treatment of patients treated with combination ivosidenib (AG-120) and nivolumab. 5) To evaluate the safety and tolerability of combination ivosidenib (AG-120) and nivolumab.

Exploratory objectives:

1. To assess the relationship between treatment response and correlative studies such as plasma and bone marrow 2-HG levels, and IDH variant allele frequency.
2. Genomic characterization by assaying specimens obtained from patients using an MDS/AML specific panel through the duration of therapy to longitudinally assess mutational burden before and during therapy, and correlating this mutational data with patient outcomes
3. Correlate exploratory biomarkers including PD-L1 expression, circulating myeloid-derived suppressor cells and interferon gamma signatures to response

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Myelodysplastic Syndrome with Excess Blast 2 (MDS-EB2) or AML according to World Health Organization (WHO) 2016 classification
* Documented IDH1 mutation within 2 months of the screening
* IDH1 mutation must be confirmed by the local laboratory during the screening period.
* Age over 18 years
* Patient must have been treated with at least 1 prior line of therapy. Hydrea is not considered as 1 line of therapy.
* Patient may have been previously treated with allogeneic transplantation if the transplant was more than 6 months ago, that the patient is not with active Graft vs. Host Disease (GVHD), and provided that the patient is not at the time of inclusion on immunosuppressant
* Eastern Cooperative Oncology Group Performance Status (ECOG PS) 0 to 2
* The patient must have recovered from toxicities of any prior treatment regimen (no CTCAE grading over 1 or return to baseline)
* Adequate hepatic and renal function:
* Hepatic Total bilirubin 1.5 x the ULN unless considered due to Gilbert's syndrome, Alanine aminotransferase (ALT) (SGPT), or aspartate aminotransferase (AST) (SGOT) 2.5 x the ULN unless considered due to organ leukemic involvement
* Renal: Serum creatinine 2 x the institutional upper limit of normal (ULN)
* The patient is able to understand and sign an informed consent form
* Females of reproductive potential and fertile males with partners who are females of reproductive potential must agree to use of 2 effective forms of contraception, one being a barrier method, or must be abstinent as part of their usual lifestyle.
* The patient is willing to participate to the study, able to adhere to the study visit schedule and other protocol procedures, and has the ability to understand and sign an inform consent form

Exclusion Criteria:

* Prior exposure to IDH targeted agents
* Prior treatment with an anti-PD-1, anti-PD-L1, anti-PD-L2 antibody, or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
* Acute Promyelocytic leukemias
* Active Central Nervous System (CNS) disease
* Participants who have received a live/ attenuated vaccine within 30 days of first treatment. Any live vaccine (ex: varicella, zoster, yellow fever, rotavirus, oral polio and measles mumps, rubella (MMR) are strictly prohibited during and for a 100 days post last treatment.
* Autoimmune disease: Patients with active, known or suspected autoimmune disease. Patients with type I diabetes mellitus, hypothyroidism only requiring hormone replacement, skin disorders (such as vitiligo, psoriasis) not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
* Medical history of Progressive multifocal leukoencephalopathy
* Patients who are unable to take PO regularly, with active gastroparesis, short gut syndrome or other malabsorption syndrome.
* Any significant medical/social condition that could limit the understanding of the study or the compliance to the protocol including but not limited to uncontrolled infection, severe or uncontrolled psychiatric illness, platelet refractoriness
* Use of strong cytochrome P-450 3A4 (CYP3A) inducers or inhibitors that cannot be safely replaced by other medications. This includes: alfentanil, aprepitant, budesonide, buspirone, conivaptan, darifenacin, darunavir, dronedarone, eletriptan, eplerenone, felodipine, indinavir, fluticasone, lopinavir, lovastatin, lurasidone, maraviroc, midazolam, nisoldipine, quetiapine, saquinavir, sildenafil, simvastatin, tolvaptan, tipranavir, triazolam, ticagrelor, vardenafil and/or the CYP2B6 substrates: bupropion, efavirenz. Posaconazole and voriconazole are not strictly prohibited, but all alternatives much be explored and use of these agents must be discussed with the Sponsor PI.
* Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days prior to the first dose of nivolumab. Corticosteroids with minimal systemic absorption (for example, topical or inhalational and adrenal replacement steroid doses > 10 mg daily prednisone or equivalent are permitted in the absence of active autoimmune disease). Use of steroids to treat toxicities acceptable is acceptable based on the local investigators standard of care).
* Prior malignancies: Any malignancy less than 1 year after end of treatment. Any malignancy presenting signs of active disease. Basal cell carcinoma and superficial cervix cancer can be included.
* History of any of the following cardiovascular conditions within 12 months of enrollment: cardiac angioplasty or stenting, myocardial infarction, unstable angina, coronary artery by-pass graft surgery, symptomatic peripheral vascular disease, class III or IV congestive heart failure, as defined by the New York Heart Association. Patients with heart-rate corrected QT interval using Fridericia's method (QTcF) >=450 msec or any other factor that increases the risk of QT prolongation or arrhythmic events (eg, heart failure, hypokalemia, family history of long QT interval syndrome). Subjects with prolonged QTcF interval in the setting of bundle branch block or pacemaker should be considered with documented consultation of a cardiologist.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
* Any known history of a positive test for hepatitis B or hepatitis C virus indicating acute or chronic infection
* Supplemental oxygen dependency or clinically significant interstitial lung disease.
* Pregnant or nursing women
* Active alcohol or drug abuse
* Patient suitable for allogeneic transplantation and with an identified allogeneic donor at the time of screening.

  1. Patients post allogeneic transplantation may be included on the trial if they are:

     1. 6 months from transplantation
     2. not actively on any immunosuppressive therapy
     3. without evidence of acute or chronic GVHD.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 168 days
  1) Overall response rate (ORR) of 60%, i.e., a 20% ORR improvement (historical control ORR = 40% with Ivosidenib[AG-120] monotherapy after 2 lines of therapy20) after 6 cycles of treatment based on MDS International Working Group 2006 criteria and AML MDS International Working group MDS/AML criteria33, 34Cumulative ORR will include complete remission (CR), morphologic complete remission with incomplete blood count recovery (CRi), CR with incomplete platelet recovery (CRp) and Partial response (PR).
Change in duration of response | 12 months
  2) In the patients who respond, Improvement in duration of response to 12 months (compared to single agent ivosidenib [AG-120] 8.2 months with ivosidenib [AG-120] monotherapy)

SECONDARY OUTCOMES:
Overall survival rate | Up to 4 years
  Overall survival will be defined from the time of treatment initiation to the time of last follow up or death. Survival with censoring patients at the time of transplantation will also be evaluated.
Progression free survival rate | Up to 4 years
  Progression free survival will be defined from the time of documentation of response to the time of relapse or death or censored at the time of last follow-up. Survival with censoring patients at the time of transplantation will also be evaluated.
Amount of Allogeneic hematopoietic stem cell transplant (HSCT) patients | 2 years
  Percentage of patients bridged to HSCT

OTHER OUTCOMES:
2-hydroxyglutarate concentration | 2 years
  To measure plasma and bone marrow 2-HG concentrations

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Prebet, PhD, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States